CLINICAL TRIAL: NCT02932891
Title: An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment With DSXS Topical Product in Patients With Atopic Dermatitis
Brief Title: An Open Label, Safety Study to Assess the Potential for Adrenal Suppression.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSXS 1502a
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSXS topical (Experimental): active treatment
  Interventions: Drug: DSXS topical

INTERVENTIONS:
Drug: DSXS topical — topical treatment
  Other Names: active

SUMMARY:
An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with DSXS in Patients with Atopic Dermatitis

DETAILED DESCRIPTION:
To evaluate the potential of DSXS topical product to suppress HPA axis function in patients with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian has signed informed consent form, which meets all criteria of current FDA regulations.

Exclusion Criteria:

* Females who are pregnant, nursing, planning to become pregnant during the duration of the study, or if of child-bearing potential and sexually active and not prepared to use appropriate contraceptive methods to avoid pregnancy

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DSXS Topical Cohort 1: active treatment
  DSXS topical: topical treatment
Period: Overall Study
Arm/Group | DSXS Topical Cohort 1
Started | 28
Completed | 24
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — HPA Suppress | 2

BASELINE CHARACTERISTICS:
Arm/Group | DSXS Topical Cohort 1
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.36 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Baseline Total BSA [Mean (Standard Deviation); unit: meters squared] | 1.61 (0.24)
Baseline IGA [Count of Participants; unit: Participants]
  Clear | 0
  Minimal | 0
  Mild | 0
  Moderate Disease | 17
  Severe Disease | 11
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI is a composite score based on the severity of four different signs of atopic dermatitis (Erythema, Induration/Papulation/Edema, Lichenification, and Excoriation rated 0 to 3 in severity) in four different areas of the body (Head/Neck, Upper Limbs, Trunk, Lower Limbs) multiplied by the percent of that specific body area affected multiplied by a weighting factor. The minimum score would be 0 and the maximum score would be 72. To be eligible for participation in this study a patient must have an EASI of at least 15 at baseline. A higher EASI value represents a more severe case of eczema.
  units on a scale | 17.64 (2.69)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in the Study With HPA Axis Suppression
Description: Hypothalamic Pituitary Adrenal (HPA) Axis Response to a stimulator
Time Frame: 29 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS Topical Cohort 1
Number analyzed (Participants) | 17
Participants
  Yes | 8
  No | 9

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | DSXS Topical Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 3/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS Topical Cohort 1 (N=28)
Nasopharyngitis (Infections and infestations) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02932891/SAP_000.pdf
  • Study Protocol (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT02932891/Prot_001.pdf